CLINICAL TRIAL: NCT02082015
Title: A Randomized, Double-Blind, Sham-Controlled, Multi-center Clinical Trial to Evaluate Efficacy and Safety of rTMS 『TMS』 for Upper Extremity Motor Function Recovery in Patients With Ischemic Stroke
Brief Title: Efficacy and Safety Study of rTMS for Upper Extremity Motor Function Recovery in Ischemic Stroke Patients
Acronym: TAMAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: DongGuk University (Other); Seoul National University Hospital (Other); REMED (Unknown)
Responsible Party: Principal Investigator, Nam-Jong Paik, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E-1308-214-002
Record Dates: First submitted 2014-03-06; First posted 2014-03-07 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Stroke; Hemiplegia
Keywords: Neuronal plasticity; Transcranial magnetic stimulation; Stroke; Upper extremity; Function; Recovery
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- true coil (Experimental): Use the true coil / Low frequency rTMS / Intensity: 100% of resting motor threshold; Location: Motor hotspot in primary motor cortex for the dominant hand; Frequency: 1Hz; Number of total stimuli: 1800; Coil orientation: tangential to scalp
  Interventions: Device: Low frequency rTMS
- sham coil (Sham Comparator): Use the sham coil / Low frequency rTMS / Intensity: 100% of resting motor threshold; Location: Motor hotspot in primary motor cortex for the dominant hand; Frequency: 1Hz; Number of total stimuli: 1800; Coil orientation: vertical to scalp
  Interventions: Device: Low frequency rTMS

INTERVENTIONS:
Device: Low frequency rTMS — Intensity: 100% of resting motor threshold; Location: Motor hotspot in primary motor cortex for the dominant hand; Frequency: 1Hz; Number of total stimuli: 1800; Coil orientation: tangential to scalp
  Other Names: TMS

SUMMARY:
The purpose of this study is to Evaluate Efficacy and Safety of rTMS 『TMS』 for Upper Extremity Motor Function Recovery in Patients with Ischemic Stroke

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) can modulate the excitability of cortex but exact efficacy and safety of rTMS is not well established.

Eighty four patients will be recruited and will be divided into two groups. Each group will receive the real rTMS or sham rTMS, respectively, over the primary motor cortex of the dominant hand. Individual subject will receive ten sessions of rTMS. Each rTMS session is low frequency (1Hz), total 1800 stimulations.

The purpose of this study is to evaluate efficacy and safety of rTMS 『TMS』 for upper extremity motor function recovery in patients with ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* 20-80 yrs old
* Radiologically confirmed ischemic stroke within 90 days
* Brunnström stage 3-5 in the affected hand (ischemic stroke-induced hemiplegic side)
* Patients received stroke treatment and on secondary prevention medication
* Written informed consent

Exclusion Criteria:

* Previous medical histories of stroke, cerebral vascular operation, seizure
* Pregnancy, Breastfeeding
* Patients with hemorrhagic stroke, traumatic brain injury
* Skin lesion in the stimulation site of scalp
* Metal implants in the body (cardiac pacemaker or aneurysm clip)
* Unable to have regular physical and occupational therapies on the affected hand

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Box and Block Test (affected hand) | up to 17 days
  Before rTMS (baseline) and 10 days after the completion of 10 sessions of rTMS

SECONDARY OUTCOMES:
Box and Block Test (Affected and unaffected hand) | up to 40 days
  Before rTMS (baseline), 10 days after the completion of 10 sessions of rTMS, 40 days after rTMS start
Barthel Index | up to 40 days
  10 days after the completion of 10 sessions of rTMS, 40 days after rTMS start
National Institutes of Health Stroke Scale | up to 40 days
  10 days after the completion of 10 sessions of rTMS, 40 days after rTMS start
Fugl-Meyer Assessment Scale | up to 40 days
  10 days after the completion of 10 sessions of rTMS, 40 days after rTMS start
Grip strength (hand grip, pinch grip, lateral prehension, three jaw chuck) | up to 40 days
  10 days after the completion of 10 sessions of rTMS, 40 days after rTMS start
Finger tapping | up to 40 days
  10 days after the completion of 10 sessions of rTMS, 40 days after rTMS start
B-stage (hand and arm) | up to 40 days
  10 days after the completion of 10 sessions of rTMS, 40 days after rTMS start
Modified Ashworth scale (wrist flexor and extensor, Elbow flexor and extensor, Long finger flexor spasticity) | up to 40 days
  10 days after the completion of 10 sessions of rTMS, 40 days after rTMS start

OTHER OUTCOMES:
Vital Sign | up to 40 days
  Before rTMS (baseline), 10 days after the completion of 10 sessions of rTMS, 40 days after rTMS start

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Jong Paik, MD, PhD, Principal Investigator — Department of Rehabilitation Medicine, Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seongnam, Korea
Locations (3):
- South Korea (3):
  - DongGuk University Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim WS, Kwon BS, Seo HG, Park J, Paik NJ. Low-Frequency Repetitive Transcranial Magnetic Stimulation Over Contralesional Motor Cortex for Motor Recovery in Subacute Ischemic Stroke: A Randomized Sham-Controlled Trial. Neurorehabil Neural Repair. 2020 Sep;34(9):856-867. doi: 10.1177/1545968320948610. Epub 2020 Aug 18. PMID 32807013